CLINICAL TRIAL: NCT05178160
Title: Lung Ultrasound-Guided PEEP Titration Versus Standard Protocol in Patients With COVID-19 ARDS Treated With CPAP: a Single Center Prospective Trial
Brief Title: Positive End Espiratory Pressure Trial in Coronavirus Disease 19 Treated With Continuous Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Maria delle Grazie Hospital (Other)
Responsible Party: Principal Investigator, Giorgio Bosso, MD, Santa Maria delle Grazie Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2N-01-COVID 19
Record Dates: First submitted 2021-12-31; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: COVID-19; PEEP trial; CPAP; lung ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): All the patients undergo to helmet-CPAP setting PEEP at 10 cmH2O and performing a blood gas analysis after 2 hours
  Interventions: Other: PEEP Standard Protocol
- Group B (Experimental): All the patients undergo to helmet-CPAP. PEEP was increased from 5 to 7.5 and 10 cmH20 in 30-minute steps during which lung ultrasound and blood gas analyses were repeated. The best PEEP was setted as the PEEP value before the appearance of lung pulse and with a PaO2/FiO2 levels stable or major than 20% in comparison to the basal value
  Interventions: Other: PEEP Standard Protocol

INTERVENTIONS:
Other: PEEP Standard Protocol — All the patients treated with CPAP receive a PEEP standard of 10 cmH2O with a fixed FiO2

SUMMARY:
Consecutive patients with hypoxemic respiratory failure, CT evidence of bilateral pneumonia and diagnosis of Coronavirus Disease 19 (COVID-19) with molecular nasopharyngeal swab consecutively admitted to the COVID Care Unit of the "Santa Maria delle Grazie" Hospital were enrolled. All the patients with clinical indication for Continuous Positive Airway Pressure (CPAP) were randomized 1:1 into two groups: Group A received a fixed Positive End Expiratory Pressure (PEEP) of 10 centimetre of water (cmH2O), Group B underwent the PEEP trial to identify the optimal PEEP (defined as the highest value that preceded the appearance of the "lung pulse" at lung ultrasound and that determined an increase in PaO2/FiO2 by at least 20%). Primary endpoint was defined as a composite in-hospital mortality+intubation, secondary endpoint was the improvement of PaO2/FiO2. As safety indicator, the incidence of pneumothorax was collected.

DETAILED DESCRIPTION:
Consecutive COVID-19 patients affected by Acute Respiratory Syndrome (ARDS) admitted to COVID Care Unit of "Santa Maria delle Grazie" Hospital, Pozzuoli (Naples, Italy), were prospectively enrolled in the study. Inclusion criteria were: age > 18 years, diagnosis of Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) infection confirmed by means of a nucleic acid test by real-time reverse transcription polymerase chain reaction (RT-PCR) on specimen from nasopharyngeal swab, bilateral interstitial pneumonia at CT scan; hypoxemic respiratory failure defined as PaO2 (partial pressure of oxygen) to FiO2 (fraction of inspired oxygen) ratio < 200.

As exclusion criteria were considered: type 2 respiratory failure; hemodynamic instability requiring vasopressors and/or inotropes support; CT evidence of pneumothorax/pneumomediastinum; concomitant acute medical disease (stroke; myocardial infarction; septic shock; gastrointestinal bleeding; acute renal failure requiring dialysis) who could affect the prognosis independent from COVID - 19.

All the patients enrolled underwent clinical history, physical examination, laboratory tests, arterial blood gas analysis, lung ultrasound, chest CT. During the hospital stay, the patients were treated according to the standard and experimental protocol available; therapies administered, and collateral effects were collected.

All participants gave their written informed consent. All the patients eligible to receive CPAP were consecutively 1:1 randomized to PEEP trial (Group A) or standard treatment (Group B).

In the Group A, PEEP was increased from 5 to 7.5 and 10 cmH20 in 30-minute steps during which lung ultrasound and blood gas analyses were repeated. PEEP responsiveness was evaluated comparing ultrasound findings and arterial blood gas parameters during oxygen supplementation with helmet-CPAP at different PEEP levels (5, 7.5 and 10, respectively), maintaining the same FiO2. A PEEP-responder is defined as a subject with clinical and/or arterial blood gases improvement with helmet-CPAP without signs of lung hyperinflation. The best PEEP was defined as the PEEP value before the appearance of lung pulse and with a PaO2/FiO2 levels stable or major than 20% in comparison to the basal value. In the Standard practice group CPAP was set at 10 cmH2O for all patients and a blood gas analysis was performed after 2 hours.

Endotracheal intubation was considered in presence of impaired respiratory mechanics, worsening of respiratory acidosis, decreased mental status.

Primary outcome was defined by a composite of hospital mortality and need of endotracheal intubation. Secondary outcome was considered the effect of CPAP on PaO2/FiO2 and respiratory rate. As a safety indicator the incidence of pneumothorax was considered.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* diagnosis of SARS-CoV-2 infection confirmed by means of RT-PCR on specimen from nasopharyngeal swab;
* bilateral interstitial pneumonia at CT scan;
* hypoxemic respiratory failure defined as PaO2/FiO2 < 200 at blood gas analyses.

Exclusion Criteria:

* type 2 respiratory failure;
* hemodynamic instability requiring vasopressors and/or inotropes support;
* CT evidence of pneumothorax/pneumomediastinum;
* concomitant acute medical disease (stroke; myocardial infarction; septic shock; gastrointestinal bleeding; acute renal failure requiring dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome | From date of randomization until the date of discharge or of endotracheal intubation or death from any cause, whichever came first, assessed up to 90 days.
  composite of hospital mortality and need of endotracheal intubation

SECONDARY OUTCOMES:
Secondary outcome | From date of randomization until the date of discharge or of endotracheal intubation or death from any cause, whichever came first, assessed up to 90 days.
  effect on P/F ratio at blood gas analyses

OTHER OUTCOMES:
Safety outcome | From date of randomization until the date of discharge or of endotracheal intubation or death from any cause, whichever came first, assessed up to 90 days.
  incidence of pneumothorax and/or pneumomediastinum

CONTACTS AND LOCATIONS:
Overall Officials: Fabio G Numis, MD, Study Chair — Santa Maria delle Grazie Hospital
Locations (1):
- COVID CARE UNIT Santa Maria delle Grazie Hospital, Pozzuoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosso G, Allegorico E, Pagano A, Porta G, Serra C, Minerva V, Mercurio V, Russo T, Altruda C, Arbo P, De Sio C, Dello Vicario F, Numis FG. Lung ultrasound as diagnostic tool for SARS-CoV-2 infection. Intern Emerg Med. 2021 Mar;16(2):471-476. doi: 10.1007/s11739-020-02512-y. Epub 2020 Oct 3. PMID 33011929
- [Result] Pagano A, Porta G, Bosso G, Allegorico E, Serra C, Dello Vicario F, Minerva V, Russo T, Altruda C, Arbo P, Mercurio V, Numis FG. Non-invasive CPAP in mild and moderate ARDS secondary to SARS-CoV-2. Respir Physiol Neurobiol. 2020 Sep;280:103489. doi: 10.1016/j.resp.2020.103489. Epub 2020 Jul 3. PMID 32629100
- [Result] Paolini V, Faverio P, Aliberti S, Messinesi G, Foti G, Sibila O, Monzani A, De Giacomi F, Stainer A, Pesci A. Positive end expiratory pressure in acute hypoxemic respiratory failure due to community acquired pneumonia: do we need a personalized approach? PeerJ. 2018 Jan 30;6:e4211. doi: 10.7717/peerj.4211. eCollection 2018. PMID 29404202